CLINICAL TRIAL: NCT04715763
Title: Randomized, Double-Blind, Placebo-Controlled Pilot Clinical Trial of the Safety and Efficacy of Telmisartan for the Treatment of COVID-19 in Hospitalized Patients
Brief Title: INvestigating TELmisartin Study
Acronym: INTEL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment due to decrease in COVID-19 rates locally
Sponsor: University of Hawaii (Other)
Collaborators: Queens Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H053
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Telmisartan

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to Telmisartan (80 mg) vs placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Telmisartan (80 mg) (Active Comparator): Telmisartan 80 mg (given as two 40 mg encapsulated tablets) given orally each day x 21 days
  Interventions: Drug: Telmisartan Oral Product
- Placebo (Placebo Comparator): Two placebo capsules given orally each day x 21 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan Oral Product — Angiotensin Receptor Blocker (ARB) FDA approved for use in hypertension and for cardiovascular risk reduction
  Other Names: Micardis
  Arms: Telmisartan (80 mg)
Drug: Placebo — Gelatin capsules filled with an inactive ingredient
  Arms: Placebo

SUMMARY:
This study will enroll 40 inpatients hospitalized for COVID-19 at Queens' Medical Center. Participants will be randomized 1:1 to Telmisartan (80 mg) vs placebo to be administered orally once daily x 21 days.

DETAILED DESCRIPTION:
The study is intended to assess, in a pilot study, the effect of telmisartan in mitigating the severity of COVID-19 related disease in hospitalized patients. Data on clinical course and lab values will be passively abstracted from Queen's standard of care evaluations on COVID-19 in-patients. Participants will be monitored closely as an outpatient if/when discharged prior to day 21. The only study-specific procedure will be a blood draw of ten (10) cc to be collected for research purposes at entry and at day 4 and day 21 of study for the evaluation of the renin-angiotensin system (RAS) system and for various blood biomarkers of organ function/coagulation, inflammation, leukocyte chemotaxis, tissue remodeling/fibrosis and immune exhaustion.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent prior to initiation of any study procedures.
* Within 72 hours of initial hospitalization for acute COVID-19 disease management
* Male or non-pregnant female adult ≥18 years of age at time of enrolment.
* Able to easily swallow pills

Exclusion Criteria:

* Systolic blood pressure less than 100 mmHg
* Self-reported history of decompensated liver failure
* Pregnancy or breast feeding
* Allergy to the study medication
* Current use of ARB, ACE inhibitors, or angiotensin receptor/neprilysin inhibitors (ARNIs). Blood pressure medications in other classes will be permitted as long as the systolic BP is >100 mmHg
* Currently receiving vasopressors for hypotension
* Prior reaction or intolerance to ARB, ACE Inhibitor or ANRI for whom study participation would not be advisable in the opinion of the study team
* Current use of and on-going need for aliskiren, lithium, digoxin, and potassium sparing diuretics such as spironolactone
* Participating in other drug clinical trials EXCEPT for other COVID-19 treatment trials which will be allowed with the permission of the Corresponding PI or Co-PI and concurrence of the treating physician/hospitalist
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 10x upper limit of normal (ULN) within 24 hours of baseline
* Absolute neutrophil count (ANC) < 1000/mL within 24 hours of baseline
* Platelet count < 50,000/mL within 24 hours of baseline.
* Patients with acute kidney injury (AKI) or chronic kidney disease (CKD) including individuals on hemodialysis may be enrolled based on the investigator's clinical judgement.
* Any serious medical condition/ abnormality or other issues that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study or suggests that the study is not in the patient's best interest
* In the opinion of the investigator, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalization | Over the 21 day period of study
  Number of days of patient's hospitalization

SECONDARY OUTCOMES:
Duration of supplemental oxygen | over the 21 days of study
  Median number of days patients required supplemental oxygen in each arm
Duration of mechanical ventilation | over the 21 days of study
  Median number of days patients required mechanical ventilation in each arm
Number of deaths | over the 21 days of study
  Total number of deaths during the study period in each arm
Number of grade 3 and greater adverse events | over the 21 days of study
  Total number of Grade 3 and greater adverse events that occurred in each arm
Clinical severity of disease | On day 4 and day 21 of study
  Clinical severity of disease as assessed by WHO Clinical Status ordinal scale (scores range from minimum value of 1 (not hospitalized, no limitations on activities) to maximum value of 7 (death); higher is worse outcome.

OTHER OUTCOMES:
Angiotensin 1-7 /Angiotensin II ratio | From entry to day 4 of study
  Change in Angiotensin 1-7/ Angiotensin II ratio

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia M Shikuma, Principal Investigator — University of Hawaii at Manoa John A Burns School of Medicine
Locations (1):
- Queen's Medical Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No